CLINICAL TRIAL: NCT01962753
Title: Depression in the Elderly and Cerebral Amyloid Plaques: Characterization by [18F] AV-45 Affectives Symptoms and Amyloïd Plaques (ASAP)
Acronym: ASAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PHRN10-VC/ ASAP
Record Dates: First submitted 2013-10-10; First posted 2013-10-14 (Estimated); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Elderly; Major Depression
Keywords: Affective symptoms as prodromal stage of Alzheimer
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 18FAV45 (Experimental)
  Interventions: Drug: 18FAV45

INTERVENTIONS:
Drug: 18FAV45 — Admnistration of 18FAV45 if patient is compliant with one of those treatment: Seroplex, Zoloft, Deroxat, Venlafaxine, Mirtazapine, Moclamine,

SUMMARY:
The primary objective of the study is to compare the brain amyloid load in fully, partially and non remitting depressed elderly patients at 8 weeks of antidepressant therapy, by using PET with [F18]AV45.

DETAILED DESCRIPTION:
The main aim of this study is to assess the brain amyloid load in treated depressed elderly subjects using PET with [F18]AV45. The investigators hypothesize that the brain amyloid load will be higher in non or partially remitting depressed subjects treated with antidepressants than in fully remitting ones. An additional two years follow-up will allow comparing the brain amyloid load at baseline between those who will have evolved towards MCI or MA and those who will not, including ApoE genotype, the cognitive performances at baseline, the hippocampus volume as assessed by MRI, the type and profile of mood disorder (number of past episodes, age at first episode, vascular risk factor profile, response profile to antidepressants), as covariates.

ELIGIBILITY:
Inclusion Criteria

* Adult 55 years or older
* Native language : french
* Study period > 7 years
* Major depression defined on the DSM-IV criteria assessed by MINI and HDRS score of 10 or over
* Affiliation to the national health insurance system
* Signed informed consent

Exclusion Criteria

* History of alcoholism or drug addiction
* MMSE less than or equal to 17
* Major depression with psychotic features
* Depressive episode resistant, patient who received two different antidepressants well conducted without significant therapeutic response
* Any current or past episode of mania, schizophrenia or any other psychotic disorder
* Any past history of stroke or Parkinson's disease
* Any current significant unstable illness
* Any past diagnosis of Alzheimer's disease
* Any current treatment by AcethylCholinesterae inhibitor, memantine or antidepressant therapy.
* Contraindications to MRI in patients with:

  1. Metallic foreign body eye.
  2. Any implanted electronic medical irremovably (pacemaker, neurostimulator, cochlear implants ...)
  3. Metal heart valve,
  4. Vascular clips formerly located on cranial aneurysm.
* Contraindications to antidepressants
* History of progressive disease that can affect the central nervous system such as uncontrolled diabetes, blood pressure greater than or equal to 180/100; chronic lung disease with hypoxia, head trauma with loss of consciousness greater than or equal to 15 minutes; brain surgery, encephalitis, recently treated cancer (<1 year), altered cerebral metabolism including subjects with stroke sequelae extended. Patients with lacunar stroke without thalamic or striatal may be included.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2012-05-10 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-01-22 (Actual)

PRIMARY OUTCOMES:
standards uptakes values (SUVr) | 2 months

SECONDARY OUTCOMES:
Residual cognitive deficits | 2 years
  The residual cognitive deficits (presence/absence) will be considered as a categorical variable.
  The ApoE genotype will also be considered as categorical variables, as well as vascular risk factor profile, WMH at MRI. MADRS, NPI and IA scores as well as the hippocampus volume will be considered as continuous variables.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent CAMUS, Principal Investigator — University Hospital of Tours
Locations (10):
- France (10):
  - University Hospital of Besançon- Jean Minjoz, Besançon
  - University Hospital of Caen, Caen
  - University Hospital of Lille, Lille
  - University Hospital of Nice, Nice
  - Sainte-Anne Hospital, Paris
  - University hospital of Rennes-Guillaume Régnier, Rennes
  - Le Rouvray Hospital, Sotteville-lès-Rouen
  - University Hospital of Strasbourg - HUS, Strasbourg
  - University Hospital of Toulouse - Purpan, Toulouse
  - University Hospital of Tours, Tours